CLINICAL TRIAL: NCT01206686
Title: Effect of Time-Slot Scheduling on Flu Vaccination Rates
Brief Title: The Effect of Time-Slot Scheduling on Flu Vaccination Rates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Harvard University (Other); Yale University (Other); Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 810589
Record Dates: First submitted 2010-09-14; First posted 2010-09-22 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Seasonal Influenza
Keywords: seasonal influenza; behavioral economics; nudge; implementations intentions; vaccination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 Hour Planning Prompt (Experimental)
  Interventions: Behavioral: Planning Prompt
- 2 Hour Planning Prompt (Experimental)
  Interventions: Behavioral: Planning Prompt
- 1 Day Planning Prompt (Experimental)
  Interventions: Behavioral: Planning Prompt
- Default Planning Prompt (Experimental)
  Interventions: Behavioral: Default Appointment
- Control (Active Comparator)
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Planning Prompt — Patients were prompted to write down a planned date (and in some cases time) for receiving a flu shot.
  Arms: 1 Day Planning Prompt; 1 Hour Planning Prompt; 2 Hour Planning Prompt
Behavioral: Default Appointment — Patients were given a suggested date and time for receiving a flu shot.
  Arms: Default Planning Prompt
Behavioral: Control — Patients were provided with basic information (present in all conditions) about when and where they could receive a flu shot, but they were given no further treatment.
  Arms: Control

SUMMARY:
The goal of this project is to see if encouraging an individual to privately choose in advance a narrow time window in which to obtain a flu vaccination shot affects the likelihood that he or she will become vaccinated.

DETAILED DESCRIPTION:
Influenza causes 36,000 U.S. deaths per year, but influenza immunization rates average just 28%. Behavioral "nudges" may increase the effectiveness of immunization reminder mailers at little or no added cost. Past psychology research has demonstrated that prompting people to form an implementation plan of the form, "When situation x arises, I will implement response y," increases attainment of desired goals because the desired behavior is linked to a concrete future moment. We study whether adding a planning prompt to a vaccination reminder mailer increases immunization rates.

ELIGIBILITY:
Inclusion Criteria:

* seasonal influenza vaccine indications according to the CDC
* employees of partner corporations executing study

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2009-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Receipt of seasonal influenza vaccination | up to 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katherine L Milkman, Ph.D., Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States